CLINICAL TRIAL: NCT00257660
Title: A Phase III Multicentre, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Dysport® for the Treatment of Cervical Dystonia
Brief Title: Randomized, Placebo-Controlled Study of AbobotulinumtoxinA (Dysport®) for the Treatment of Cervical Dystonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-47-52120-051; 2005-000709-70 (EudraCT Number)
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Results first posted 2010-05-10 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Drug: abobotulinumtoxinA (Dysport®)
  Interventions: Biological: Botulinum toxin type A
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — 500 units
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: 1
Drug: Placebo — 500 units
  Arms: 2

SUMMARY:
The aim of this study is to demonstrate the effectiveness and safety of 500 units of Dysport manufactured at a new manufacturing facility in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Cervical dystonia with at least 18 months since onset, and previously untreated with botulinum toxin or previously treated with botulinum toxin type A or B with a minimum interval of 16 weeks since the last injection and having returned at least to their usual pre-treatment status
* TWSTRS severity, disability and total scores meeting the defined criteria at baseline

Exclusion Criteria:

* Pure anterocollis or pure retrocollis
* In apparent remission from cervical dystonia
* Previous poor response to the last two botulinum toxin type A or type B treatments
* Being treated with type B toxin due to lack of efficacy to type A toxin or have known neutralizing antibodies to type A toxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2005-10-10 (Actual); Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (22):
- United States (18):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - USC School of Medicine, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Wayne State University Medical Center, Southfield, Michigan
  - Albany Medical Center, Albany, New York
  - Beth Israel Medical Center, New York, New York
  - Columbia University, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Allegeheny General, Pittsburgh, Pennsylvania
  - University of Texas Southwest, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Swedish Neuroscience, Seattle, Washington
- Russia (4):
  - Scientific Research Institute of Neurology, RAMS, Moscow
  - Clinic "Cecil Plus", Moscow
  - Municipal Multi-Speciality Hospital #2, Saint Petersburg
  - St Petersburg Pavlov State Medical University, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Result] Truong D, Brodsky M, Lew M, Brashear A, Jankovic J, Molho E, Orlova O, Timerbaeva S; Global Dysport Cervical Dystonia Study Group. Long-term efficacy and safety of botulinum toxin type A (Dysport) in cervical dystonia. Parkinsonism Relat Disord. 2010 Jun;16(5):316-23. doi: 10.1016/j.parkreldis.2010.03.002. Epub 2010 Mar 31. PMID 20359934
- [Derived] Mordin M, Masaquel C, Abbott C, Copley-Merriman C. Factors affecting the health-related quality of life of patients with cervical dystonia and impact of treatment with abobotulinumtoxinA (Dysport): results from a randomised, double-blind, placebo-controlled study. BMJ Open. 2014 Oct 16;4(10):e005150. doi: 10.1136/bmjopen-2014-005150. PMID 25324317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 16 centres in the USA and 4 centres in Russia from October 2005 until September 2006
Groups:
- Dysport 500 Units; Placebo: Single intramuscular injection into the clinically indicated neck muscles in a single dosing session wherever possible
Period: Overall Study
Arm/Group | Dysport 500 Units | Placebo
Started | 55 | 61
Completed | 45 | 38
Not Completed | 10 | 23
Not completed — Lack of Efficacy | 5 | 23
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — PI & Subject Schedule Conflicts | 1 | 0
Not completed — No longer wanted to do blood draws | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dysport 500 Units | Placebo | Total
Number analyzed (Participants) | 55 | 61 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 50 | 96
  >=65 years | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (13.4) | 53.9 (12.5) | 53.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 18 | 23 | 41
Region of Enrollment [Number; unit: participants]
  United States | 41 | 47 | 88
  Russian Federation | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)
Description: TWSTRS is comprised of three different components which are severity, disability & pain. There is an ordinal scale for each component and the score range for each is the following: for severity from 0 (absence of severity) to 35 (max severity), for disability from 0 (no disability) to 30 (max disability) and for pain from 0 (no pain) to 20 (max pain). TWSTRS total score is the sum of the 3 component scores, with a range from 0 to a maximum of 85. The change in TWSTRS total score is the score at week 4 minus the score at baseline.
Time Frame: Baseline and Week 4
Population: The analysis was performed on the intention to treat population which consisted of 55 subjects receiving Dysport and 61 Placebo. There were 4 subjects for Dysport and 3 for placebo who were not assessed on TWSTRS score at Week 4. As there was no imputation of missing TWSTRS score values, these 7 subjects were not taken into account.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 51 | 58
points on a scale
  Change in TWSTRS total score | -13.99 (12.33) | -5.23 (9.33)
  Baseline TWSTRS total score | 43.83 (7.97) | 45.81 (8.78)
  Week 4 TWSTRS total score | 30.04 (12.65) | 40.22 (11.75)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — A hierarchical testing procedure was applied for the primary and secondary outcome measures ranked in the order of priority listed. At each step of the hierarchical testing procedure, there was one comparison and p<0.05 was considered significant; Treatment group, baseline TWSTRS score, center and previous treatment by botulinum toxin or not were fitted in the ANCOVA model; Mean Difference (Net) = -8.84, 95% CI 2-sided [-12.94 to -4.74] — Baseline TWSTRS total scores are analysed for all subjects of ITT population, while the analysis at Week 4 excludes the scores for the 7 subjects who were not assessed. Mean difference = difference in adjusted least squares mean (Dysport - Placebo)

2. Secondary Outcome: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)
Description: as for outcome 1
Time Frame: Baseline and Week 8
Population: The analysis was performed on the intention to treat population which consisted of 55 subjects receiving Dysport and 61 Placebo. There were 9 subjects for Dysport and 15 for placebo who were not assessed on TWSTRS score at Week 8. As there was no imputation of missing TWSTRS score values, these 24 subjects were not taken into account.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 46 | 46
points on a scale
  Change in TWSTRS total score | -13.82 (11.53) | -5.59 (11.37)
  Baseline TWSTRS total score | 43.83 (7.97) | 45.81 (8.78)
  Week 8 TWSTRS total score | 29.31 (10.99) | 39.64 (13.50)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -8.81, 95% CI [-12.91 to -4.71] — Baseline TWSTRS total scores are analysed for all subjects of ITT population, while the Week 8 analysis excludes the scores for the 24 subjects who were not assessed. Mean difference = difference in adjusted least squares mean (Dysport - Placebo)

3. Secondary Outcome: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Total Score
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: The analysis was performed on the intention to treat population which consisted of 55 subjects receiving Dysport and 61 Placebo. There were 10 subjects for Dysport and 17 for placebo who were not assessed on TWSTRS score at Week 12. As there was no imputation of missing TWSTRS score values, these 27 subjects were not taken into account.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 45 | 44
points on a scale
  Change in TWSTRS total score | -6.98 (11.12) | -4.53 (7.75)
  Baseline TWSTRS total score | 43.83 (7.97) | 45.81 (8.78)
  Week 12 TWSTRS total score | 36.04 (11.76) | 40.76 (11.08)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p = 0.019, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -4.12, 95% CI [-7.55 to -0.68] — Baseline TWSTRS total scores are analysed for all subjects of ITT population, while the Week 12 analysis excludes the scores for the 27 subjects who were not assessed. Mean difference = difference in adjusted least squares mean (Dysport - Placebo)

4. Secondary Outcome: Subject Visual Analogue Score (VAS) for Cervical Dystonia (CD) Symptom Assessment
Description: The assessment was a continuous 100 mm horizonal line with a scale of 0 mm (no symptoms)to 100 mm (worst possible symptoms).
Time Frame: Baseline and Week 4
Population: Analysis was performed on intention to treat population which consisted of 55 subjects on Dysport and 61 on Placebo. There were 5 subjects on Dysport and 8 on placebo who were not assessed on the change in subject VAS score for CD symptoms at Week 4. There was no imputation of missing VAS scores, so these 13 subjects were not taken into account.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 50 | 53
points on a scale
  Change in Subject VAS for CD symptoms | -24.2 (29.5) | -6.7 (20.8)
  Baseline Subject VAS for CD symptoms | 67.7 (19.7) | 63.6 (18.9)
  Week 4 Subject VAS for CD symptoms | 44.3 (24.4) | 55.7 (20.6)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Treatment group, baseline Subject VAS symptom score, center and previous treatment by botulinum toxin or not were fitted in the ANCOVA model; Mean Difference (Net) = -15.2, 95% CI [-24.0 to -6.4] — Analysis at baseline (and on change at Week 4) excludes 4 subjects (and 13 subjects respectively) of ITT population who were not assessed. Mean difference=difference in adjusted least squares mean (Dysport-placebo)

5. Secondary Outcome: Investigator VAS for CD Symptom Assessment
Description: as for outcome 4
Time Frame: Baseline and Week 4
Population: Analysis was performed on intention to treat population which consisted of 55 subjects receiving Dysport and 61 Placebo. There were 3 subjects for Dysport and 5 for placebo who were not assessed on the change in investigator VAS score at Week 4. As there was no imputation of missing VAS scores, these 8 subjects were not taken into account.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 52 | 56
points on a scale
  Change in Investigator VAS for CD symptoms | -23.1 (22.1) | -9.1 (20.2)
  Baseline Investigator VAS for CD symptoms | 62.3 (15.8) | 65.3 (18.0)
  Week 4 Investigator VAS for CD symptoms | 40.3 (21.7) | 56.8 (21.8)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Treatment group, baseline Investigator VAS CD symptom score, center and previous treatment by botulinum toxin or not were fitted in the ANCOVA model; Mean Difference (Net) = -14.2, 95% CI [-22.3 to -6.1] — Analysis at baseline (and on change at Week 4) excludes 3 subjects (and 8 subjects respectively) of ITT population who were not assessed. Mean difference=difference in adjusted least squares mean (Dysport-placebo)

6. Secondary Outcome: Subject VAS for CD Symptom Assessment
Description: The assessment was a continuous 100 mm horizonal line with a scale of 0 mm (no symptoms)to 100mm (worst possible symptoms).
Time Frame: Baseline and Week 8
Population: Analysis was performed on intention to treat population which consisted of 55 subjects on Dysport and 61 on Placebo. Missing assessments at Week 8 were imputed using Last Observation Carried Forward (LOCF) methodology. There was no imputation for 4 patients on placebo with missing baseline and Week 4 values.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 55 | 57
points on a scale
  Change in subject VAS for CD symptoms | -24.6 (30.0) | -5.4 (25.4)
  Baseline subject VAS for CD symptoms | 67.7 (19.7) | 63.6 (18.9)
  Week 8 subject VAS for CD symptoms | 44.7 (24.9) | 57.8 (27.5)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Treatment group, baseline Subject VAS Pain score, center and previous treatment by botulinum toxin or not were fitted in the ANCOVA model; Mean Difference (Net) = -16.95, 95% CI [-25.8 to -8.1] — Analysis at baseline (and on change at Week 8) excludes 4 subjects (and 4 subjects respectively) of ITT population who were not assessed. Mean difference=difference in adjusted least squares mean (Dysport-placebo)

7. Secondary Outcome: Investigator's VAS for CD Symptom Assessment
Description: as for outcome 4
Time Frame: Baseline and week 8
Population: Analysis was performed on intention to treat population which consisted of 55 subjects on Dysport and 61 on Placebo. Missing assessments at Week 8 were imputed using Last Observation Carried Forward (LOCF) methodology. There was no imputation for 3 patients with missing baseline and Week 4 values.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 54 | 59
points on a scale
  Change in Investigator VAS for CD symptoms | -20.5 (22.7) | -5.0 (21.3)
  Baseline Investigator VAS for CD symptoms | 62.3 (15.8) | 65.3 (18.0)
  Week 8 Investigator VAS for CD symptoms | 40.8 (22.3) | 60.8 (24.6)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Treatment group, baseline Investigator VAS Pain score, center and previous treatment by botulinum toxin or not were fitted in the ANCOVA model; Mean Difference (Net) = -16.0, 95% CI [-24.2 to -7.8] — Analysis at baseline (and on change at Week 8) excludes 3 subjects (and 3 subjects respectively) of ITT population who were not assessed. Mean difference=difference in adjusted least squares mean (Dysport-placebo)

8. Secondary Outcome: Subject VAS for CD Symptom Assessment
Description: as for outcome 4
Time Frame: Baseline and week 12
Population: Analysis was performed on intention to treat population which consisted of 55 subjects on Dysport and 61 on Placebo. Missing assessments at Week 12 were imputed using Last Observation Carried Forward (LOCF) methodology. There was no imputation for 4 patients on placebo with missing baseline, Week 4 and Week 8 values.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 55 | 57
points on a scale
  Change in subject VAS for CD symptoms | -14.4 (25.2) | -4.6 (23.3)
  Baseline subject VAS for CD symptoms | 67.7 (19.7) | 63.6 (18.9)
  Week 12 subject VAS for CD symptoms | 55.4 (25.5) | 58.2 (25.7)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 6, analysis 1]; Mean Difference (Net) = -11.05, 95% CI [-19.0 to -3.1] — Analysis at baseline (and on change at Week 12) excludes 4 subjects (and 4 subjects respectively) of ITT population who were not assessed. Mean difference=difference in adjusted least squares mean (Dysport-placebo)

9. Secondary Outcome: Investigator's VAS for CD Symptom Assessment
Description: The assessment was a continuous 100 mm horizonal line with a scale of 0 mm (no symptoms) to 100 mm (worst possible symptoms).
Time Frame: Baseline and week 12
Population: Analysis was performed on intention to treat population which consisted of 55 subjects on Dysport and 61 on Placebo. Missing assessments at Week 12 were imputed using Last Observation Carried Forward (LOCF) methodology. There was no imputation for 3 patients with missing baseline, Week 4 and Week 8 values.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 54 | 59
points on a scale
  Change in Investigator VAS for CD symptoms | -8.5 (18.9) | -5.8 (15.8)
  Baseline Investigator VAS for CD symptoms | 62.3 (15.8) | 65.3 (18.0)
  Week 12 Investigator VAS for CD symptoms | 54.8 (20.8) | 60.0 (21.5)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p = 0.028, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 7, analysis 1]; Mean Difference (Net) = -7.05, 95% CI [-13.3 to -0.8] — Analysis at baseline (and on change at Week 12) excludes 3 subjects (and 3 subjects respectively) of ITT population who were not assessed. Mean difference=difference in adjusted least squares mean (Dysport-placebo)

10. Secondary Outcome: SF-36 Mental Health Summary Score
Description: SF-36 is a Quality of Life scale comprising eight individual domains. The QoL score for each domain is on a scale from 0 (worst health possible) to 100 (best health possible). SF-36 Mental Health Summary Score is derived from four individual domains (vitality, social functioning, role limitations due to emotional problems and mental health).
Time Frame: Week 8
Population: Analysis was performed on intention to treat population which consisted of 55 subjects on Dysport and 61 on Placebo. There were 13 subjects on Dysport and 24 on placebo who were not assessed on the change in mental health summary at Week 8. There was no imputation of missing scores, so these 37 subjects were not taken into account.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 42 | 37
points on a scale
  Change in SF-36 Mental health summary Score | 4.11 (9.18) | 2.48 (8.12)
  Baseline SF-36 Mental health summary Score | 44.52 (10.41) | 43.31 (11.14)
  Week 8 SF-36 Mental health summary Score | 49.00 (8.69) | 43.41 (12.30)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p = 0.061, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Treatment group, baseline SF-36 mental health summary score, center and previous treatment by botulinum toxin or not were fitted in the ANCOVA model; Mean Difference (Net) = 3.65, 95% CI [-0.17 to 7.47] — Analysis at baseline (and on change at Week 8) excludes 3 subjects (and 37 subjects respectively) of ITT population who were not assessed. Mean difference=difference in adjusted least squares mean (Dysport-placebo)

11. Secondary Outcome: SF-36 Physical Health Summary Score
Description: SF-36 is a Quality of Life scale comprising eight individual domains. The QoL score for each domain is on a scale from 0 (worst health possible) to 100 (best health possible). SF-36 Physical Health Summary Score is derived from four individual domains (physical functioning, role physical, bodily pain and general health).
Time Frame: Week 8
Population: Analysis was performed on intention to treat population which consisted of 55 subjects on Dysport and 61 on Placebo. There were 13 subjects on Dysport and 24 on placebo who were not assessed on the change in physical health summary at Week 8. There was no imputation of missing scores, so these 37 subjects were not taken into account.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 42 | 37
points on a scale
  Change in SF-36 Physical health summary score | 4.37 (5.46) | -0.64 (6.41)
  Baseline SF-36 Physical health summary score | 39.42 (8.84) | 43.18 (7.89)
  Week 8 SF-36 Physical health summary score | 43.70 (8.76) | 42.49 (8.84)
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Treatment group, baseline SF-36 physical health summary score, center and previous treatment by botulinum toxin or not were fitted in ANCOVA model; Mean Difference (Net) = 4.66, 95% CI [1.73 to 7.58] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Number of Participants Considered by the Investigator to be Overall Treatment Successes
Description: The number of participants considered to be overall treatment successes by the investigator at week 12 was assessed.
Time Frame: Week 12
Population: Analysis was performed on intention to treat population which consisted of 55 participants on Dysport and 61 on Placebo.
Measure: Number; unit: participants
Arm/Group | Dysport 500 Units | Placebo
Number analyzed (Participants) | 55 | 61
participants | 32 | 10
Statistical Analysis 1: Comparison: Dysport 500 Units vs Placebo; The number of participants considered treatment successes was analysed using a logistic model with treatment, strata (naive or non-naive) and center as factors in the model; Test type: Superiority or Other; p < 0.0001, odds ratio — [p-value comment as in outcome 1, analysis 1]; The odds ratio represents the odds of success on Dysport versus Placebo stratified for strata and country; Odds Ratio (OR) = 7.206, 95% CI [3.01 to 17.26]

ADVERSE EVENTS:
Arm/Group | Dysport 500 Units | Placebo
Serious Adverse Events (participants affected / at risk) | 0/55 | 1/61
Other Adverse Events (participants affected / at risk) | 11/55 | 5/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport 500 Units (N=55) | Placebo (N=61)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport 500 Units (N=55) | Placebo (N=61)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 0 (0)
Injection site pain (General disorders) | 3 (3) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A publication of results from all sites in this multicenter study is expected. If the sponsor no longer plans this or 6 months after study completion at all sites, the PI may publish the results. He will supply any proposed publication to the sponsor for review and comment at least 30 days before submission for publication. If the sponsor believes a patent application should be filed, the publication will be delayed for another 60 days or until patent filing; with a maximum delay of 90 days.